CLINICAL TRIAL: NCT03583424
Title: A Phase I/II Trial of Venetoclax and BEAM Conditioning Followed by Autologous Stem Cell Transplantation for Patients With Primary Refractory Non-Hodgkin Lymphoma
Brief Title: Venetoclax, Carmustine, Etoposide, Cytarabine, and Melphalan Before Stem Cell Transplant in Treating Participants With Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Kami Maddocks, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-17225; NCI-2018-01039 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic Cell Transplantation Recipient; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory Marginal Zone Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Transformed Indolent Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin | interventions — Carmustine; carmustine, poliferprosan 20 drug combination; Cytarabine; Etoposide; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Melphalan; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, BEAM) (Experimental): Participants receive venetoclax PO QD on days -10 to -1, carmustine IV on day -6, etoposide IV BID on days -5 to -2, cytarabine IV BID on days -5 to -2, and melphalan IV on day -1. Participants then undergo hematopoietic cell transplantation on day 0.
  Interventions: Drug: Carmustine; Drug: Cytarabine; Drug: Etoposide; Procedure: Hematopoietic Cell Transplantation; Drug: Melphalan; Drug: Venetoclax

INTERVENTIONS:
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Procedure: Hematopoietic Cell Transplantation — Undergo hematopoietic cell transplantation
  Other Names: HCT; Hematopoietic Stem Cell Transplantation; HSCT; stem cell transplantation
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta

SUMMARY:
This phase I/II trial studies the side effects and best dose of venetoclax when given together with carmustine, etoposide, cytarabine, and melphalan before stem cell transplant in treating participants with non-Hodgkin lymphoma that has come back or does not respond to treatment. Drugs used in chemotherapy, such as venetoclax, carmustine, etoposide, cytarabine, and melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before a stem cell transplant helps kill any cancer cells that are in the body and helps make room in the patient?s bone marrow for new blood-forming cells (stem cells) to grow.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of venetoclax that can be safely combined with carmustine, etoposide, cytarabine, and melphalan (BEAM) prior to autologous stem cell transplant which will the recommended phase II dose (RP2D).

II. Determine the safety and efficacy of venetoclax as measured by overall response rate (ORR) at day 100, 12-month survival and freedom from relapse (FFR-12).

SECONDARY OBJECTIVES:

I. Long term effects (progression-free survival [PFS] and overall survival [OS]) of addition of venetoclax to BEAM.

II. Correlation of response and survival with expression of BCL-2, BCL-XL, and MCL-1 as measured by immunohistochemistry (IHC).

OUTLINE: This is a dose-escalation study of venetoclax.

Participants receive venetoclax orally (PO) once daily (QD) on days -10 to -1, carmustine intravenously (IV) on day -6, etoposide IV twice daily (BID) on days -5 to -2, cytarabine IV BID on days -5 to -2, and melphalan IV on day -1. Participants then undergo hematopoietic stem cell transplantation on day 0.

After completion of study treatment, participants are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed diagnosis of non-Hodgkin?s lymphoma that has relapsed, or is refractory, after upfront induction therapy. Excluded histologies are T-cell lymphomas, post-transplant lymphoproliferative disorder, Burkitt lymphoma, lymphoblastic lymphoma, chronic lymphocytic leukemia/small lymphocytic lymphoma. All other histologies are eligible that include but not limited to: diffuse-large B-cell lymphoma, follicular lymphoma (grades I, II, and III), marginal zone lymphoma, transformed indolent lymphoma, grey zone lymphoma, and undifferentiated B-cell lymphoma. Patients with non-Hodgkin's lymphoma (NHL) who are at high risk of relapse can be enrolled in sustained partial response (PR) after induction chemotherapy (PR1)
* Expected survival of more than six months
* Karnofsky performance status >= 80%
* Within 1 week prior to initiation of treatment: Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 3 x upper limits of normal (ULN) unless due to disease
* Within 1 week prior to initiation of treatment: Total bilirubin < 2 x ULN unless due to disease
* Within 1 week prior to initiation of treatment: Calculated glomerular filtration rate (GFR) 30 ml/min
* Within 1 week prior to initiation of treatment: Absolute neutrophil count (ANC) > 500 cells/mm^3
* Within 1 week prior to initiation of treatment: Platelet count > 50 mm^3
* Left ventricular ejection fraction >= 40%
* Diffusion capacity of carbon monoxide (DLCO) >= 50% predicted
* Ability to collect 2 x 10^6/kg CD34+ cells for transplantation
* Patient must be otherwise eligible for autologous stem cell transplantation (ASCT) per local institutional guidelines
* No serious disease, or condition, that, in the opinion of the investigator, would compromise the patient?s ability to participate in the study
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subjects who sustained a complete metabolic response (CMR) by positron emission tomography (PET)-computed tomography (CT) (Deauville score of =< 3) after salvage chemotherapy unless lymphoma relapsed less than 12 months from the first day of last cycle of induction chemotherapy OR patient required more than 2 lines of salvage chemotherapy to sustain a CMR
* Subjects receiving any other investigational agents
* Prior treatment with venetoclax
* Patients with central nervous system (CNS) involved by lymphoma can be included if CNS disease is deemed controlled prior to enrollment as determined by the investigator. Patients with uncontrolled CNS disease will be excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to venetoclax or other agents used in this study
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are human immunodeficiency virus (HIV) positive and receiving combination antiretroviral therapy will be excluded; because of the potential for pharmacokinetic interactions with venetoclax
* Female patients who are pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women. Male or female patients, who are sexually active and of the child bearing age, must be willing to practice accepted birth control measures

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kami Maddocks, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For this study, dose level 3 was determined to be the maximum tolerated dose (MTD). Therefore, 10 patients who were accrued for the expansion phase were treated at the MTD. Combining with 3 patients treated at dose level 3 in the escalation phase, all 13 patients were treated at the same dose level. Therefore, they were grouped together for the results reporting.
Groups:
- Cohort A (Venetoclax 400 mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation; Cohort B (Venetoclax 800mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation); Cohort C (Venetoclax 1200mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation): Participants receive Venetoclax PO QD on days -10 to -1, carmustine IV on day -6, etoposide IV BID on days -5 to -2, cytarabine IV BID on days -5 to -2, and melphalan IV on day -1. Participants then undergo hematopoietic cell transplantation on day 0.
  Carmustine: Given IV
  Cytarabine: Given IV
  Etoposide: Given IV
  Hematopoietic Cell Transplantation: Undergo hematopoietic cell transplantation
  Melphalan: Given IV
  Venetoclax: Given PO
Period: Overall Study
Arm/Group | Cohort A (Venetoclax 400 mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation | Cohort B (Venetoclax 800mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation) | Cohort C (Venetoclax 1200mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation)
Started | 3 | 3 | 13
Completed | 3 | 3 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: For this study, dose level 3 was determined to be the maximum tolerated dose (MTD). Therefore, 10 patients who were accrued for the expansion phase were treated at the MTD. Combining with 3 patients treated at dose level 3 in the escalation phase, all 13 patients were treated at the same dose level. Therefore, they were grouped together for the results reporting.
Groups:
- Cohort A (Venetoclax 400mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation); Cohort B (Venetoclax 800mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation); Cohort C (Venetoclax 1200mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation): Participants receive Venetoclax PO QD on days -10 to -1, carmustine IV on day -6, etoposide IV BID on days -5 to -2, cytarabine IV BID on days -5 to -2, and melphalan IV on day -1. Participants then undergo hematopoietic cell transplantation on day 0.
  Carmustine: Given IV
  Cytarabine: Given IV
  Etoposide: Given IV
  Hematopoietic Cell Transplantation: Undergo hematopoietic cell transplantation
  Melphalan: Given IV
  Venetoclax: Given PO
- Total: Total of all reporting groups
Arm/Group | Cohort A (Venetoclax 400mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation) | Cohort B (Venetoclax 800mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation) | Cohort C (Venetoclax 1200mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation) | Total
Number analyzed (Participants) | 3 | 3 | 13 | 19
Age, Continuous [Median (Full Range); unit: years] | 64 [55 to 69] | 52 [49 to 64] | 61 [41 to 72] | 61 [41 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 4
  Male | 3 | 2 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 13 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 3 | 2 | 13 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 13 | 19

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Venetoclax Defined to be the Dose Cohort Below Which 3 Out of 6 Patients Experience Dose Limiting Toxicities or the Highest Dose Cohort of 1200 mg, if 2 Dose Limiting Toxicities Are Not Observed at Any Dose Cohort
Time Frame: Up to 2 years
Measure: Number; unit: mg
Arm/Group | Treatment (Venetoclax, BEAM)
Number analyzed (Participants) | 10
mg | 1200

2. Primary Outcome: Overall Response Rate
Description: Will be estimated as the proportions of patients who achieve a complete response or partial response divided by the number of evaluable patients. Each will be reported with their associated 95% confidence interval.
Time Frame: At day 100
Measure: Number; unit: percentage of participants
Groups:
- Cohort B (Venetoclax 800 mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation; Cohort C (Venetoclax 1200 mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation: Participants receive venetoclax PO QD on days -10 to -1, carmustine IV on day -6, etoposide IV BID on days -5 to -2, cytarabine IV BID on days -5 to -2, and melphalan IV on day -1. Participants then undergo hematopoietic cell transplantation on day 0.
  Carmustine: Given IV
  Cytarabine: Given IV
  Etoposide: Given IV
  Hematopoietic Cell Transplantation: Undergo hematopoietic cell transplantation
  Melphalan: Given IV
  Venetoclax: Given PO
Arm/Group | Cohort A (Venetoclax 400 mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation | Cohort B (Venetoclax 800 mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation | Cohort C (Venetoclax 1200 mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation
Number analyzed (Participants) | 3 | 3 | 13
percentage of participants | 33 | 67 | 69

3. Secondary Outcome: Number of Participants With Progression of Disease
Description: Estimated using Kaplan-Meier method.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A (Venetoclax 400mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation; Cohort B (Venetoclax 800mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation); Cohort C (Venetoclax 1200mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation): Participants receive Venetoclax PO QD on days -10 to -1, carmustine IV on day -6, etoposide IV BID on days -5 to -2, cytarabine IV BID on days -5 to -2, and melphalan IV on day -1. Participants then undergo hematopoietic cell transplantation on day 0.
  Carmustine: Given IV
  Cytarabine: Given IV
  Etoposide: Given IV
  Hematopoietic Cell Transplantation: Undergo hematopoietic cell transplantation
  Melphalan: Given IV
  Venetoclax: Given PO
Arm/Group | Cohort A (Venetoclax 400mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation | Cohort B (Venetoclax 800mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation) | Cohort C (Venetoclax 1200mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation)
Number analyzed (Participants) | 3 | 3 | 13
Participants | 3 | 0 | 5

4. Secondary Outcome: Number of Participants Free From Relapse
Description: Estimated using Kaplan-Meier method.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B (Venetoclax 800mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation; Cohort C (Venetoclax 1200mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation: Participants receive venetoclax PO QD on days -10 to -1, carmustine IV on day -6, etoposide IV BID on days -5 to -2, cytarabine IV BID on days -5 to -2, and melphalan IV on day -1. Participants then undergo hematopoietic cell transplantation on day 0.
  Carmustine: Given IV
  Cytarabine: Given IV
  Etoposide: Given IV
  Hematopoietic Cell Transplantation: Undergo hematopoietic cell transplantation
  Melphalan: Given IV
  Venetoclax: Given PO
Arm/Group | Cohort A (Venetoclax 400mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation | Cohort B (Venetoclax 800mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation | Cohort C (Venetoclax 1200mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation
Number analyzed (Participants) | 3 | 3 | 13
Participants | 0 | 3 | 6

5. Secondary Outcome: Overall Survival
Description: Estimated using Kaplan-Meier method.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A (Venetoclax 400mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation | Cohort B (Venetoclax 800mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation | Cohort C (Venetoclax 1200mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation
Number analyzed (Participants) | 3 | 3 | 13
Months | NA [NA to NA] — Median Overall Survival not reached | NA [NA to NA] — Median Overall Survival not reached | NA [NA to NA] — Median Overall Survival not reached

ADVERSE EVENTS:
Time Frame: The National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting for up to 2 years
Arm/Group | Cohort A (Venetoclax 400mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation | Cohort B (Venetoclax 800mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation | Cohort C (Venetoclax 1200mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 4/13
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Venetoclax 400mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation (N=3) | Cohort B (Venetoclax 800mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation (N=3) | Cohort C (Venetoclax 1200mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation (N=13)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 4 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Venetoclax 400mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation (N=3) | Cohort B (Venetoclax 800mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation (N=3) | Cohort C (Venetoclax 1200mg and BEAM Conditioning Followed by Autologous Stem Cell Transplantation (N=13)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder, GI (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (at line site) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT03583424/Prot_SAP_000.pdf